CLINICAL TRIAL: NCT05922891
Title: Effectiveness of Tezepelumab on Asthma Control and Cough: A Prospective, Multi-center, Observational Study
Brief Title: Tezepelumab PRO Study
Acronym: TezepelumabPRO
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00025
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study assesses the impact of tezepelumab treatment not only on asthma control but also on cough specific Health-Related Quality of Life (HRQoL). Asthma control can be evaluated using Asthma Control Questionnaire (ACQ). Cough symptom which is one of the symptoms related airway hyperresponsiveness can be assessed via the relevant questionnaire, Leicester Cough Questionnaire (LCQ). There is moderate negative correlation between ACQ and LCQ . Improvements in both asthma control and cough symptom by tezepelumab would clarify effectiveness of Tezepelumab in real-world. Though Tezepelumab is recently approved in Japan, there is no real-world evidence on tezepelumab, particularly on above mentioned symptoms.

Thus, this study aims to estimate effectiveness of tezepelumab on asthma and cough symptoms in real world settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years who provide informed consent and who receive new prescription of Tezepelumab as per the physician's decision at baseline according to the package insert saying "Tezepelumab is given to patient with asthma (limited to severe or refractory patient whose asthma symptoms cannot be controlled even with existing treatment)"
2. ACQ-6 ≥1.5 at baseline
3. Patients with persistent cough ≥8 weeks up until the baseline visit according to The Japanese Respiratory Society Guidelines for the Management of Cough and Sputum 2019

Exclusion Criteria:

1. Patients who had asthma exacerbation within one month before study enrollment
2. Patients who had the biologics treatment in following period prior to the enrollment

   * omalizumab in 2 or 4 weeks depending on the body weight and total IgE amount
   * mepolizumab in 4 weeks
   * Benralizumab in 8 weeks
   * Dupilumab in 2 weeks
3. Patients with cough related diseases other than asthma as determined by treating physicians
4. Patients participating in studies that affect this study (study with other interventional treatment to evaluate efficacy/safety of treatment in patients with cough, asthma, or allergic/eosinophilic diseases)
5. Any disorder, including heart failure, malignancy, morbid obesity(BMI≧35) , respiratory infectious disease that is not stable (e.g. patients who need medical treatment) in the opinion of the investigator and could:

   * Affect the safety of the patient throughout the study
   * Impede the patient's ability to complete the entire duration of study
6. Patients with pregnancy or lactation period

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a total of 90 patients with severe uncontrolled asthma who initiate new prescription of tezepelumab.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Mean change in ACQ-6 at week 52 from baseline | Baseline and Week 52
  To estimate change of asthma control as measured by the ACQ-6 in patients who initiated Tezepelumab at week 52 from baseline

SECONDARY OUTCOMES:
Mean change in LCQ at week 52 from baseline | Baseline and Week 52
  To estimate change of cough-specific health-related quality of life in patients who initiated Tezepelumab at week 52 from baseline
Mean change in LCQ at week 4, 12, 24 from baseline | Baseline, Week 4, Week 12 and Week 24
  To estimate change of cough-specific health-related quality of life in patients who initiated Tezepelumab at week 4, 12, 24 from baseline
Mean change in ACQ-6 at week 4, 12, 24 from baseline | Baseline, Week 4, Week 12 and Week 24
  To estimate change of asthma control as measured by the ACQ-6 in patients who initiated Tezepelumab at week 4, 12, 24 from baseline
Asthma exacerbation rate during 52 weeks before/after Tezepelumab initiation Ratio of annual asthma exacerbation rate between previous 52 weeks and Tezepelumab treated 52 weeks | During 52 weeks before/after Tezepelumab initiation
  To estimate asthma exacerbation during 52 weeks before/after Tezepelumab initiation

CONTACTS AND LOCATIONS:
Locations (29):
- Japan (29):
  - Research Site, Aomori
  - Research Site, Bunkyō City
  - Research Site, Fujisawa
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Hamamatsu
  - Research Site, Hiroshima
  - Research Site, Iizuka
  - Research Site, Izumo
  - Research Site, Kawasaki
  - Research Site, Kitakyushu
  - Research Site, Kiyose
  - Research Site, Kurashiki
  - Research Site, Matsusaka
  - Research Site, Minami
  - Research Site, Minato
  - Research Site, Nagoya
  - Research Site, Naka
  - Research Site, Niigata
  - Research Site, Nishinomiya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shinagawa City
  - Research Site, Shinjuku
  - Research Site, Shizuoka
  - Research Site, tabashi City
  - Research Site, Tennōjichō-kita
  - Research Site, Ube
  - Research Site, Yonago

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials/studies via the request portal. All request will be evaluated as per the AZdisclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home